CLINICAL TRIAL: NCT01797120
Title: Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Fulvestrant (Faslodex) Plus Everolimus in Post-Menopausal Patients With Hormone-Receptor Positive Metastatic Breast Cancer Resistant to Aromatase Inhibitor Therapy
Brief Title: Study of Fulvestrant +/- Everolimus in Post-Menopausal, Hormone-Receptor + Metastatic Breast Ca Resistant to AI
Acronym: PrE0102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PrE0102
Record Dates: First submitted 2013-02-14; First posted 2013-02-22 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Post-Menopausal Patients; Hormone-Receptor Positive; Resistant to Aromatase Inhibitor Therapy; Fulvestrant; Faslodex; mTOR Inhibitor; Everolimus; RAD001; Afinitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Everolimus; Sirolimus; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fulvestrant & Everolimus (Active Comparator): Fulvestrant Day 1 & 15 of Cycle 1, then Day 1 of all subsequent cycles (every 28 days for 12 cycles) plus everolimus daily x 12 cycles.
  Interventions: Drug: Fulvestrant; Drug: Everolimus
- Fulvestrant & Placebo (Placebo Comparator): Fulvestrant Day 1 & 15 of Cycle 1, then Day 1 of all subsequent cycles (every 28 days for 12 cycles) plus placebo daily x 12 cycles.
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant 500 mg Day 1 & 15 of Cycle 1, then 500 mg Day 1 of all subsequent cycles (every 28 days for 12 cycles).
  If no evidence of disease progression after 12 cycles, unblind and continue same dose and schedule until progression or unacceptable toxicity.
  Other Names: Faslodex
Drug: Everolimus — Everolimus 10 mg (2 tablets) daily x 12 cycles.
  If no evidence of disease progression after 12 cycles, unblind and continue same dose and schedule until progression or unacceptable toxicity.
  Other Names: mTOR Inhibitor; RAD001; Afinitor
  Arms: Fulvestrant & Everolimus
Drug: Placebo — Placebo for Everolimus (2 tablets) daily x 12 cycles. Placebo manufactured to mimic everolimus tablet.
  Other Names: Sugar Pill
  Arms: Fulvestrant & Placebo

SUMMARY:
Post-menopausal women with hormone-receptor positive (HR+) metastatic breast cancer resistant to aromatase inhibitor (AI) therapy will be randomized to receive Fulvestrant (Faslodex) with Everolimus or Fulvestrant (Faslodex) with a placebo (no active ingredients).

Fulvestrant has demonstrated activity when used as first, second, or third line endocrine therapy, making it an attractive therapy for combination with other agents. In addition, it is commonly reserved for use following disease progression on AI therapy.

Everolimus is an orally administered drug that blocks a signaling pathway called "mTOR". "mTOR" acts as a regulator for many processes in the body, including cell growth. Blocking this pathway may have an effect on cell growth.

The combination of a novel class of agents (mTOR inhibitors) and an established standard treatment for metastatic HR+ breast cancer may potentially increase the clinical benefit by targeting multiple different biological pathways.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed malignancy in women worldwide. In the United States, an estimated 230,480 new cases of invasive breast cancer were diagnosed in 2011, with 39,520 breast cancer deaths. In 40-80% of women with node-positive disease at diagnosis, their breast cancer will recur. When distant metastases occur, median survival is 18 to 36 months from time of recurrence. Among the 60-70% of women with HR+ breast cancer, 40-60% of them will benefit from endocrine therapy. Endocrine therapy has shown to yield similar survival rates in hormone-sensitive disease as compared to chemotherapy; although response rates are lower and responses develop more slowly. Endocrine therapy is considerably less toxic than chemotherapy, and is therefore the preferred treatment option for patients with HR+ disease.

Endocrine therapy represents the foundation of treatment for HR+ metastatic and locally advanced breast cancer. Multiple compounds in varying classes exist, and those most widely used include the selective estrogen receptor modulators (SERMs), aromatase inhibitors (AIs), and the selective estrogen receptor down-regulators (SERDs). Although the utility of these drugs is well established, as many as 50% of women with HR+ breast cancer will fail to respond to endocrine treatment. Moreover, those who do respond will inevitably develop acquired resistance.

Fulvestrant is the first drug which acts as a pure estrogen receptor (ER) antagonist without known agonist effects. It competitively binds to the ERs with an approximately 100 times greater affinity than that of tamoxifen. Fulvestrant promotes the degradation of ERs and subsequently prevents ER-mediated gene transcription.

Everolimus (RAD001) is an oral derivative of rapamycin that is an m-TOR inhibitor. At cellular and molecular levels, everolimus acts as a signal transduction inhibitor. Everolimus selectively inhibits mTOR (mammalian target of rapamycin); a key and highly conserved serine-threonine kinase which is present in all cells and is a central regulator of protein synthesis and ultimately cell growth, cell proliferation, angiogenesis and cell survival. mTOR is the only currently known target of everolimus.

In oncology, everolimus has been in clinical development since 2002 for patients with various hematologic and non-hematologic malignancies as a single agent or in combination with antitumor agents, including cytotoxic chemotherapeutic agents, targeted therapies, antibodies and hormonal agents.

Patients will be randomized (1:1) to receive everolimus or placebo with fulvestrant after consideration of stratification factors of performance status (0 vs. 1), measurable disease (yes vs. no), and prior chemotherapy for metastatic disease (yes vs. no).

Patients will be evaluated for disease response every 12 weeks, and treated until disease progression or unacceptable toxicity or withdrawal of consent for a maximum of 12 cycles (48 weeks).

Patients with no evidence of progressive disease who remain on study after completing 12 cycles are unblinded and continue to receive fulvestrant alone (if originally randomized to placebo) or in combination with everolimus (if originally randomized to everolimus) at the same dose and schedule. Patients will continue to be evaluated for disease response every 12 weeks and continue until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. ≥18 years.
3. ECOG Performance Status 0 or 1.
4. Histologically or cytologically confirmed adenocarcinoma of the breast.
5. Stage IV disease or inoperable locally advanced disease.
6. ER and/or PR-positive disease. Tumors must be HER-2/neu negative or equivocal.
7. Aromatase Inhibitor (AI) resistant, defined as:

   * relapsed while receiving adjuvant therapy with an AI or,
   * progressive disease while receiving an AI for metastatic disease
8. Received one prior cycle of fulvestrant within 28 days of randomization are eligible.

   * ≥2 prior doses of fulvestrant are not eligible
9. Must be female and postmenopausal.
10. May have received ≤1 prior systemic chemotherapy regimen for metastatic disease.
11. Adequate organ function:

    * Whole Blood Cells (WBC) ≥3.0 x 10⁹/L, Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L and platelet count ≥100 x 10⁹/L
    * hemoglobin ≥9 g/dL
    * serum bilirubin ≤1.5 X ULN (Upper Limit of Normal)
    * Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≤2.5 X ULN (≤5 x ULN in patients with liver metastases)
    * serum creatinine ≤1.5 X ULN
    * serum albumin ≥3 g/dL
    * fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5 x ULN.
    * Prothrombin time (PT) with international normalized ratio (INR) ≤1.5
12. May have measurable disease, non-measurable disease, or both.
13. Basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix within the past five years treated with curative intent. History of prior malignancy are eligible if disease-free for >3 years.

Exclusion Criteria:

1. Major surgery or significant traumatic injury within 4 weeks of randomization or patients that may require major surgery during the course of the study.
2. Investigational agents within 4 weeks of randomization.
3. Anticancer treatment within 4 weeks of randomization, with the following exceptions:

   * Bisphosphonates or Zometa for bone metastases
   * a GnRH analog is permitted if the patient had progressive disease on a GnRH (Gonadotropin-Releasing Hormone) analog plus a SERM (Selective Estrogen Receptor Modulators) or an AI; the GnRH analog may continue but the SERM or AI must be discontinued.
4. Prior treatment with an mTOR inhibitor.
5. Receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent ≥ 5 mg prednisone or equivalent daily.
6. Receive immunization with attenuated live vaccines within one week of randomization or during the study period.
7. Current or a prior history of brain metastases or leptomeningeal disease. Must not have rapidly progressive, life-threatening metastases.
8. Known hypersensitivity/history of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus or fulvestrant.
9. Congenital or acquired immune deficiency at increased risk of infection.
10. Impairment of gastrointestinal function/disease that may significantly alter the absorption of everolimus.
11. Active, bleeding diathesis.
12. History of any condition or uncontrolled intercurrent illness that in the opinion of the local investigator might interfere with or limit the patient's ability to comply with the protocol or pose additional or unacceptable risk to the patient.
13. Severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    * Symptomatic congestive heart failure of New York Heart Association Class III or IV
    * Unstable angina pectoris, myocardial infarction within 6 months of randomization, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
    * History of symptomatic pulmonary disease or non-malignant pulmonary disease requiring treatment.
    * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
    * Active (acute or chronic) or uncontrolled severe infections
    * Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh Class C).

Note: Detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah S Kornblum, MD, Study Chair — Saint Barnabas Cancer Center, Montefiore Medical Center
Locations (25):
- United States (25):
  - Marin Cancer Care, Greenbrae, California
  - Stanford University, Stanford, California
  - SwedishAmerican Regional Cancer Center, Rockford, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - St. Joseph Mercy Hospital (MI Cancer Consortium), Ann Arbor, Michigan
  - Metro MN, Saint Louis Park, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Beth Israel, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Toledo COP, Toledo, Ohio
  - Hematology & Oncology Associates of Northeastern PA, PC, Dunmore, Pennsylvania
  - Penn State University, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh- Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital- McGlinn Family Regional Cancer Center, West Reading, Pennsylvania
  - Main Line Heath System, Wynnewood, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Health System, La Crosse, Wisconsin
  - ProHealth Care Inc. (Waukesha), Waukesha, Wisconsin
  - Aurora Cancer Care, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Result] Kornblum N, Zhao F, Manola J, Klein P, Ramaswamy B, Brufsky A, Stella PJ, Burnette B, Telli M, Makower DF, Cheema P, Truica CI, Wolff AC, Soori GS, Haley B, Wassenaar TR, Goldstein LJ, Miller KD, Sparano JA. Randomized Phase II Trial of Fulvestrant Plus Everolimus or Placebo in Postmenopausal Women With Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Metastatic Breast Cancer Resistant to Aromatase Inhibitor Therapy: Results of PrE0102. J Clin Oncol. 2018 Jun 1;36(16):1556-1563. doi: 10.1200/JCO.2017.76.9331. Epub 2018 Apr 17. PMID 29664714
- See also: Fulvestrant Plus Everolimus or Placebo in Postmenopausal Women With ER-Positive Metastatic Breast Cancer Resistant to Aromatase Inhibitor — http://www.ncbi.nlm.nih.gov/pubmed/29664714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 131 patients were enrolled from 23 institutions between May 2013 and November 2015.
Groups:
- Fulvestrant & Everolimus: Fulvestrant Day 1 & 15 of Cycle 1, then Day 1 of all subsequent cycles (every 28 days for 12 cycles) plus everolimus daily x 12 cycles.
  Fulvestrant: Fulvestrant 500 mg Day 1 & 15 of Cycle 1, then 500 mg Day 1 of all subsequent cycles (every 28 days for 12 cycles).
  If no evidence of disease progression after 12 cycles, unblind and continue same dose and schedule until progression or unacceptable toxicity.
  Everolimus: Everolimus 10 mg (2 tablets) daily x 12 cycles.
  If no evidence of disease progression after 12 cycles, unblind and continue same dose and schedule until progression or unacceptable toxicity.
- Fulvestrant & Placebo: Fulvestrant Day 1 & 15 of Cycle 1, then Day 1 of all subsequent cycles (every 28 days for 12 cycles) plus placebo daily x 12 cycles.
  Fulvestrant: Fulvestrant 500 mg Day 1 & 15 of Cycle 1, then 500 mg Day 1 of all subsequent cycles (every 28 days for 12 cycles).
  If no evidence of disease progression after 12 cycles, unblind and continue same dose and schedule until progression or unacceptable toxicity.
  Placebo: Placebo for Everolimus (2 tablets) daily x 12 cycles. Placebo manufactured to mimic everolimus tablet.
Period: Overall Study
Arm/Group | Fulvestrant & Everolimus | Fulvestrant & Placebo
Started | 66 | 65
Completed | 0 | 0
Not Completed | 66 | 65
Not completed — Disesae progression | 37 | 49
Not completed — Adverse Event | 13 | 5
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Symptomatic progression | 2 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Physician Decision | 3 | 0
Not completed — still on treatment | 2 | 4
Not completed — never start protocol therapy | 2 | 0

BASELINE CHARACTERISTICS:
Population: all randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant & Everolimus | Fulvestrant & Placebo | Total
Number analyzed (Participants) | 66 | 65 | 131
Age, Continuous [Median (Full Range); unit: years] | 64 [39 to 92] | 59 [35 to 85] | 63 [35 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 131
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 56 | 49 | 105
  Black | 8 | 11 | 19
  Others | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival documented by Physical Exam, CT Scan or MRI in post-menopausal patients with hormone-receptor positive metastatic breast cancer that is resistant to aromatase inhibitor therapy treated with fulvestrant and everolimus compared to fulvestrant alone from randomization to documented disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 3 months until progression or up to 3 years
Population: all randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant & Everolimus | Fulvestrant & Placebo
Number analyzed (Participants) | 66 | 65
months | 10.3 [7.6 to 13.8] | 5.1 [3.0 to 8.0]
Statistical Analysis 1: Comparison: Fulvestrant & Everolimus vs Fulvestrant & Placebo; Test type: Superiority; p = 0.02, Log Rank; Log rank test was stratified on ECOG performance status, measurable disease, and prior chemotherapy for metastatic disease; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.40 to 0.92]

2. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is defined as number of patients with objective response (complete response or partial response) or stable disease for at least 24 weeks divided by number of patients randomized in each arm. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR) is defined as >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease; Complete Response (CR) is defined as disappearance of all target lesions.
Time Frame: Every 3 months until progression or up to 3 years
Population: all randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Fulvestrant & Everolimus | Fulvestrant & Placebo
Number analyzed (Participants) | 66 | 65
proportion of patients | 0.636 [0.509 to 0.751] | 0.415 [0.294 to 0.544]
Statistical Analysis 1: Comparison: Fulvestrant & Everolimus vs Fulvestrant & Placebo; Test type: Superiority; p = 0.01, Fisher Exact

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as number of patients with complete or partial response (by Physical Exam, CT or MRI) divided by number of patients randomized in each arm
Time Frame: Every 3 months until progression or up to 3 years
Population: all randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Fulvestrant & Everolimus | Fulvestrant & Placebo
Number analyzed (Participants) | 66 | 65
proportion of patients | 0.182 [0.098 to 0.296] | 0.123 [0.055 to 0.228]
Statistical Analysis 1: Comparison: Fulvestrant & Everolimus vs Fulvestrant & Placebo; Test type: Superiority; p = 0.47, Fisher Exact

4. Secondary Outcome: Overall Survival
Description: Overall survival will be characterized using Kaplan-Meier plots and other descriptive metrics.
Time Frame: Every 3 months until progression or up to 3 years
Population: all randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant & Everolimus | Fulvestrant & Placebo
Number analyzed (Participants) | 66 | 65
months | 28.3 [19.5 to 29.6] | 31.4 [21.8 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment

ADVERSE EVENTS:
Time Frame: Assessed at the end of each cycle (1 cycle=4 weeks) while on treatment and 30 days after the last dose of protocol therapy. Treatment continued for a maximum of 48 weeks (12 cycles) in the absence of disease progression, unacceptable toxicity or withdrawal of consent.
Description: All-cause mortality is the death rate among all patients, rather than in patients who received at least one dose of protocol therapy and reported toxicity data.
Arm/Group | Fulvestrant & Everolimus | Fulvestrant & Placebo
All-Cause Mortality (participants affected / at risk) | 30/66 | 21/65
Serious Adverse Events (participants affected / at risk) | 31/64 | 5/65
Other Adverse Events (participants affected / at risk) | 59/64 | 38/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant & Everolimus (N=64) | Fulvestrant & Placebo (N=65)
Oral mucositis (Gastrointestinal disorders) | 7 | 0
Fatigue (General disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Elevated AST (Hepatobiliary disorders) | 2 | 1
Lymphocytopenia (Blood and lymphatic system disorders) | 2 | 0
Elevated ALT (Hepatobiliary disorders) | 1 | 0
Esophageal Candidiasis (Infections and infestations) | 1 | 0
Esophagitis (Infections and infestations) | 1 | 0
Hypertension (Blood and lymphatic system disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Inflammation (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and Medical Procedures (Surgical and medical procedures) | 1 | 0
Thromboembolic Event (Cardiac disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant & Everolimus (N=64) | Fulvestrant & Placebo (N=65)
Oral mucositis (Gastrointestinal disorders) | 26 | 8
Fatigue (General disorders) | 23 | 11
Rash (Skin and subcutaneous tissue disorders) | 23 | 3
Anorexia (Gastrointestinal disorders) | 22 | 4
Anemia (Blood and lymphatic system disorders) | 18 | 3
Nausea (Gastrointestinal disorders) | 16 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 1
Diarrhea (Gastrointestinal disorders) | 13 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 10 | 2
Weight loss (General disorders) | 9 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 0
Dysgeusia (Gastrointestinal disorders) | 8 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Chills (General disorders) | 7 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 2
Vomitting (Gastrointestinal disorders) | 7 | 3
Headache (General disorders) | 6 | 6
Hot flashes (Cardiac disorders) | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
AST increased (Hepatobiliary disorders) | 4 | 1
ALT increased (Hepatobiliary disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 4 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 12 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 1
Insomnia (Gastrointestinal disorders) | 4 | 0
White blood cell decreased (Blood and lymphatic system disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-01-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT01797120/Prot_000.pdf
  • Statistical Analysis Plan (2014-03-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT01797120/SAP_001.pdf